CLINICAL TRIAL: NCT05428475
Title: Implementation and Evaluation of Improved Access to Medical Imaging for Geriatric Patients of The Royal Ottawa Hospital
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tim Lau (Other)
Collaborators: McGill University (Other)
Responsible Party: Sponsor-Investigator, Tim Lau, Clinical Lead, Geriatric Psychiatry Inpatient Unit, The Royal Ottawa Mental Health Centre
Organization: The Royal Ottawa Mental Health Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021040
Record Dates: First submitted 2022-06-10; First posted 2022-06-23 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Dementia; Cognitive Impairment; Dementia With Lewy Bodies
Keywords: The Royal; FDG-PET Imaging
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Lewy Body Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [18F]FDG-PET Scan (Experimental): Participants with unclear symptoms of cognitive impairment who will undergo the [18F]FDG-PET scan (185 MBq of [18F]FDG administered once during study).
  Interventions: Diagnostic Test: [18F]FDG-PET Scan

INTERVENTIONS:
Diagnostic Test: [18F]FDG-PET Scan — 185 MBq of [18F]FDG will be administered IV 30 minutes prior to PET scan. Images will be acquired for 30 minutes. Resulting images will be evaluated for patterns of FDG-uptake to support the diagnosis of the participant symptoms of cognitive impairment.

SUMMARY:
In this study, the investigators implement FDG-PET imaging for clients in the Geriatric Psychiatry department at The Royal Ottawa Hospital (ROH) and evaluate the impact of this advanced imaging technique on client care. This study is intended to provide supporting evidence for the continued use of FDG-PET imaging at the ROH BIC as a diagnostic support for the differential diagnosis of unclear dementia.

DETAILED DESCRIPTION:
OVERVIEW

The investigators will recruit 15 participants in the Geriatric Psychiatry department at the Royal Ottawa Hospital (ROH) who have an unclear diagnosis of dementia and their study partners. Each participant will have four study visits expected to take less than six months of involvement in total. The study partner is required to accompany the participant for all visits.

Visit 1: Informed consent and completion of pre-imaging questionnaires. Visit 2: Eligible participants undergo an FDG-PET scan at the Brain Imaging Centre (BIC).

Visit 3: Meeting with referring physician to review FDG-PET results. Visit 4: Completion of post-imaging questionnaires.

Wherever possible, Visits 1, 2 and 4 will be scheduled to coincide with regular clinical appointments. For participants who do not have decisional capacity, assent will be sought at each visit and recorded on the Continuing Consent/Assent study document. The study procedures will be described at a level that is understandable to the participant. This may mean describing one step at a time and seeking assent for that piece of the study in the moment. Both verbal and physical cues as well as feedback from the study partner will be used to support assent.

Visit 1: Eligibility Screening and Informed Consent

The first visit will begin by explaining the study procedures, reviewing the inclusion and exclusion criteria, and obtaining an informed consent. This visit will be conducted at the Royal's Geriatric Psychiatry department. Medical history, including previous diagnostic tests, current medications, current possible diagnoses and family history will be gathered from the electronic health records, the participant and/or their SDM, and the referring physician. Demographic information including age and sex will be noted. An MRI safety pre-screening will be completed to check for any contraindications to being in the MRI environment. The participant (if able) and study partner will complete a pre-scan survey (Participant Pre-Scan Survey, Study Partner Pre-Scan Survey) and the self-rated/study partner rated version of the Alzheimer's Disease Cooperative Study - Clinician's Global Impression of Change (ADCS-CGIC) (Schneider, 2006). The study partner will also be asked to complete the Mild Behavioural Impairment Checklist (MBI-C).

Visit 2: PET-MRI Scanning

Within two weeks prior to the PET-MRI scan the participant's referring physician will be required to complete a pre-scan survey. This survey must be completed prior to the PET-MRI scan visit. In this Referring Physician Pre-PET Survey, the referring physician will provide information on their diagnostic certainty via the Referring Physician Pre-PET Survey. The physician will be asked to list the diagnosis/diagnoses they are considering, based on the information they currently have, to explain the participant's symptoms of cognitive impairment. For each diagnosis, the physician is required to indicate their level of confidence in that diagnosis as a percentage, where 1% indicates complete uncertainty and 100% represents absolute certainty that the diagnosis is accurate. The physician will also provide information on the participant's current management plan related to their symptoms of cognitive impairment and attach a list of the participant's current medications. Finally, the physician will answer questions about their level of comfort and understanding of the use of FDG-PET to support the differential diagnosis of dementia symptoms.

This visit will be scheduled approximately 2 weeks after obtaining informed consent. Scheduling of this visit will be done in conjunction with the Geriatric Psychiatry department to facilitate the participant's needs and minimize the impact on the unit's workflow. The participant's study partner's schedule will also be considered.

The study partner will be required to attend the PET-MRI appointment to provide support and to observe the process. The participant must arrive fasted (no food for a minimum of 6-hours prior, only water to drink). Upon arrival at the BIC, the participant will be re-screened for any MRI and PET safety counter indications by a PET/MRI Technologist. If the study partner is not the SDM, the SDM will need to be available by phone to review the MRI and PET safety information with the PET/MRI Technologist. A blood glucose measurement (requires a small finger prick) will be taken to ensure that there is minimal competition between the PET tracer and glucose circulating in the bloodstream. This measurement will be repeated immediately before and after the scan. Prior to positioning in the scanner the participant will be injected with the PET tracer by a PET Technologist (18F-fluorodeoxyglucose, 185MBq±10%), followed by a 30-minute period of quiet rest (dark room, eyes open) to allow for tracer uptake. The client will then be positioned in the PET-MRI scanner (Siemens Biograph mMR) and at 30-minutes post-injection PET data will be acquired for 30 minutes. Simultaneously, a structural anatomical image (T1) will be acquired to allow for correction of attenuation in the PET data and to provide context for the PET images.

A neuromelanin MRI (NM-MRI) scan will be conducted to measure dopamine function. NM is a dark pigment synthesized via iron dependent oxidation of dopamine; it accumulates progressively over the lifespan. Using a non-invasive technique known as neuromelanin-sensitive magnetic resonance imaging (NM-MRI), we can measure changes in NM signal over time and ultimately how dopamine functions in the brain. NM-MRI is currently included in multiple protocols at ROH including a longitudinal study looking at this measure over the life-span in healthy controls. Dr. Cliff Cassidy, a co-investigator on this study, is a leader in the development of this technique (Cassidy, 2019). NM-MRI is a brief non-invasive MRI sequence that takes 8-minutes to acquire, and from the participant perspective is no different to the acquisition of the anatomical T1 MRI data. In this study, NM-MRI results will be compared to a database of healthy aging to explore whether NM-MRI reflects the cognitive health of the participant and has the potential to be used as a diagnostic tool.

Clinical MRI sequences may also be acquired during this time for participants who are expected to have difficulty tolerating the imaging procedure. All MRI scans will fit within the 30 minute PET acquisition time. All participants will be instructed to relax with eyes open or closed and limit head motion. A vacuum pillow is used to create padding for additional movement restriction. Earplugs will be used to reduce scanner noise. Following the PET-MRI scan the participant will be encouraged to use the washroom to reduce the radiation dose from tracer accumulated in the bladder. Following the FDG-PET scan the participant (if able) and study partner will be asked to complete a survey about their experience in the BIC. This can be completed before they leave the BIC, or done at home and returned via email/mail.

Visit 3: Review of FDG-PET Imaging Results

After the FDG-PET scan is complete the participant's images and medical history will be reviewed and a research interpretation will be provided to the participant's referring physician. It will be at the referring physician's discretion how they share these results with the participant, study partner and SDM (e.g. in person, over the phone, via Zoom) and how they use this information in the differential diagnosis of the participant.

After this visit the referring physician will be asked to complete a post-scan survey indicating any changes in diagnostic thinking and care of the patient. In this Referring Physician Post-PET Survey, the physician will repeat the exercise of listing the diagnosis/diagnoses they are considering and indicating their level of confidence in that diagnosis. Using this data we will evaluate whether physician diagnostic confidence increased with the inclusion of the FDG-PET data in the participant's workup. The physician will also provide information on any changes to the participant's management plan and attach a list of the participant's current medications. Physicians will also comment on their comfort level in using FDG-PET, whether they would order this test again, and whether they would recommend this test to other physicians.

Visit 4: 3-Month Follow-Up

Three months after Visit 3 the participant (if able), study partner and referring physician will be asked to complete a post-scan survey. The physician provides information on any additional changes made to the participant's management plan where the FDG-PET results were a contributing factor in making the change. This is done using the Referring Physician 3-Months Post-PET Survey. The participant (if able) and study partner asked to rate the importance of access to FDG-PET for other patients with similar symptom profiles using the Participant or Study-Partner 3-Month Post-PET Survey. Additionally, the participant (if completed at Visit 1) and study partner will be asked to complete the ADCS-CGIC.

DATA ANALYSIS

FDG-PET images will be reviewed by Dr. Soucy who will provide a research interpretation of the FDG-PET data. Dr. Soucy has extensive experience in the review and evaluation of FDG-PET for dementia applications. It will be clearly communicated to the referring physician that integration of the research interpretation in diagnosis and treatment (and the participant's medical records) will be at their discretion. Structural MRI data (T1) will be used in the calculation of the FDG-PET attenuation correction, and to support evaluation of the FDG-PET data by providing anatomical context.

Fully de-identified data, including the clinical data and PET data, will be shared with Dr. Jean-Paul Soucy (MD, Nuclear Medicine and Director, PET Unit, McConnell Brain Imaging Centre, Montreal Neurological Institute) at McGill University for review and generation of a research report. De-identified clinical data, contained in a password protected file, will be transferred via email to Dr. Soucy. De-identified imaging data will be transferred via the BIC's internal secure data download portal. The data transferred will be labelled by patient codes to maintain the anonymity of the participants.

Fully de-identified T1 and NM-MRI data, clinical data, and MBI-C, will be shared with Dr. Cliff Cassidy, a co-investigator on this study. Dr. Cassidy will compare the participant's data against a pre-existing database of healthy control data to evaluate whether NM-MRI has the potential to provide any additional diagnostic information in the diagnosis of the participant's symptoms.

Results from the physician surveys will be compiled to understand any changes in diagnostic thinking and therapeutic planning resulting from access to FDG-PET imaging. Participant and study partner surveys will be tabulated to highlight perceived changes in participant wellbeing and care resulting from access to FDG-PET imaging. Due to the small sample size, basic statistical tests will be used to determine the significance of changes in diagnosis and diagnostic certainty.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are able to speak and read English.
2. Participant or their Substitute Decision Maker (SDM) are able to provide written informed consent to participate in the study.
3. Participants are able to comply with the requirements of the study.
4. Participant has a study partner who will provide written informed consent to participate, is in frequent contact with the participant, will accompany the participant to FDG-PET study visit and will complete pre-/post-FDG-PET surveys.
5. Participant has a diagnosis of a cognitive impairment.
6. Participant has undergone a standard baseline clinical evaluation.
7. Participant has undergone clinical structural brain imaging (MRI or CT).
8. Structural brain imaging excluded an anatomical cause of the symptoms of cognitive impairment.
9. Participant has been evaluated by a cognitive disorders specialist.
10. Participant has an unclear underlying pathological process despite the above evaluations and the referring physician feels added clarity in the diagnosis has the potential to help with clinical management.

Exclusion Criteria:

1. Participant is not able to comply with the requirements of the study (including fasting for 6 hours, lying still in a supine position for 50 minutes).
2. Participant an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth that cannot be safely removed.
3. Participant has any contraindication to MRI or PET imaging.
4. Participant has active malignancies. This is due to the high likelihood that the participant is or will be undergoing radiation therapy.
5. Participant been exposed to other sources of radiation within the past year, where these bring their total radiation dose above the annual maximum.
6. Female participants who are pregnant or breastfeeding. All female participants of childbearing potential will be required to have a negative urine pregnancy test on the day of the FDG-PET scan. Women are considered to be of childbearing potential if they are not permanently sterile or postmenopausal (12 consecutive months with no menses without an alternative medical cause).
7. Participant has any other condition that, in the opinion of the investigator, could create a hazard to the participant's safety, endanger the study procedures, or interfere with the interpretation of study results.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Determine changes in clinician confidence in their differential diagnosis of clients with unclear symptoms of dementia. | At participation initiation for baseline measurement, 1 month, and 3 months
  The study will measure clinician diagnostic confidence pre- and post- FDG-PET using the Referring Physician Pre-PET Survey and Referring Physician Post-PET Survey.
Determine changes in Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) | At participation initiation for baseline measurement and 3 months
  The number of participants for whom a change in treatment plan occurred due to the added information from the FDG-PET scan, as reported on the Referring Physician Pre- and Post-PET Surveys, will be measured. Additionally, participant and study partner reported global impression of change over the course of the study will be tabulated to determine if any overall clinical improvement was observed (ADCS-CGIC).
  On the ADCS-CGIC, global severity at baseline scored from 1 (normal, not at all ill) to 7 (among the most extremely ill patients); and global change at follow-up scored from 1 (marked improvement) to 7 (marked worsening), where 4 indicates no change.
Identify changes in client treatment regiment as a result of access to FDG-PET imaging. | At participation initiation for baseline measurement and 3 months
  Dichotomy measure of if the treatment regiment for the client was changed (success=1) or not changed (fail=0) as a result from the FDG-PET results.
Determine participant perceptions of access to medical imaging for patients of The Royal. | At participation initiation for baseline measurement and 3 months
  Participants and their study partners will be asked about whether access to medical imaging affected their confidence in their treatment and diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Lau, MD, FRCP(C), Principal Investigator — The Royal Ottawa Hospital

IPD SHARING:
Plan to Share IPD: No